CLINICAL TRIAL: NCT04368039
Title: Normobaric Oxygen Therapy for Individuals With First-Episode Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicholas Breitborde (Other)
Responsible Party: Sponsor-Investigator, Nicholas Breitborde, Principal Investigator, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019H0424
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Psychosis; Schizophrenia; First-episode Psychosis
Keywords: psychosis; treatment; normobaric hyperoxia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Normobaric Oxygen Therapy (40% FiO2) (Experimental): 4 weeks of nightly normobaric oxygen therapy (40% FiO2)
  Interventions: Device: Normobaric Oxygen
- Placebo Condition (Placebo Comparator): 4 weeks of a placebo condition utilizing room air oxygen levels (21% FiO2)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Normobaric Oxygen — 40% FiO2 for 4 weeks
  Arms: Normobaric Oxygen Therapy (40% FiO2)
Device: Placebo — 21% FiO2 for 4 weeks
  Arms: Placebo Condition

SUMMARY:
Single-blind, randomized controlled trial of normobaric oxygen therapy among individuals with first-episode psychosis: Effects on symptomatology and cognition.

DETAILED DESCRIPTION:
Functional deficits in prefrontal, limbic, and temporal regions of the brain are well-documented among individuals with psychotic disorders. Mitochondrial dysfunction may contribute to such pathology, and effective functioning of mitochondrial activity in the brain in dependent on a sufficient supply of oxygen. These data suggest that oxygen therapy may improve symptoms in individuals with psychosis. This small pilot study will test this hypothesis.

Individuals with first-episode psychosis will be randomized to receive either (i) 4 weeks of nightly normobaric oxygen therapy (40% FiO2) or (ii) 4 weeks of a placebo condition utilizing room air oxygen levels (21% FiO2). Participants will be blinded to what condition they receive. Both conditions will be delivered via nasal cannula connected to oxygen concentrators at five liters per minute (lpm), and participants will be instructed to complete the intervention overnight while sleeping. At the end of the 4 week period, all individuals will receive an additional 4 weeks of unblinded (i.e., "open label") nightly normobaric oxygen therapy (40% FiO2). Study assessments will be completed at (i) enrollment; (ii) 4 weeks after enrollment, and (iii) 8 weeks after enrollment.

ELIGIBILITY:
* Diagnosis of a schizophrenia-spectrum disorder or mood disorder with psychotic features as determined using the Structured Clinical Interview for the DSM-5.
* Less than 5 years since the onset of frank psychotic symptoms as determined using the Symptom Onset in Schizophrenia Inventory .
* No evidence of a pre-existing intellectual disability defined as a premorbid IQ >70 as estimated using the Reading subtest of the Wide Range Achievement Test-4.
* Ages 15-35
* Non-smoker for past six months
* Absence of suicidal ideation or behavior over the past month as assessed by the Columbia Suicide Severity Rating Scale
* The American Association for Respiratory Care notes that "no absolute contraindications to oxygen therapy exist when indications [for oxygen therapy] are present."

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2025-12-07 (Estimated); Study Completion 2025-12-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cognitive functioning | 4 weeks
  Change in scores on the MATRICS Consensus Cognitive Battery (MCCB).
Change from baseline in quality of life | 4 weeks
  Change in scores on WHO Quality of Life Scale Brief (WHOQOL-BREF.
Change from baseline in social functioning | 4 weeks
  Change in scores on the Global Functioning: Social Scale. Scores on this measure range from 1-10 with higher scores indicating greater social functioning
Change from baseline in role functioning | 4 weeks
  Change in scores on the Global Functioning: Role Scale. Scores on this measure range from 1-10 with higher scores indicative of greater role functioning.
Change from baseline in health-related quality of life | 4 weeks
  Change in scores on the RAND 36-Item Health Survey.

SECONDARY OUTCOMES:
Change from baseline in suicidality | 4 weeks
  Change in occurrence in suicidal thoughts or behaviors as assessed using the Columbia Suicide Severity Rating Scale. This is a categorical rating scale that identifies the presence or absence of specific levels of severity of suicidal ideation and behavior.
Change from baseline in substance use severity | 4 weeks
  Change in scores on the HABITS scale. This scale assesses the absolute values of use of specific substances (e.g., number of cigarettes smoked)
Change from baseline in service utilization | 4 weeks
  Change in scores on the Modified Service Use and Resources Form for Schizophrenia
Change in Sleep | 4 weeks
  Change in scores on the Pittsburgh Sleep Quality Index.
Change from baseline in medication adherence | 4 weeks
  Change in scores on the Medication Adherence rating Scale. Scores on this scale range from 0-10 with higher scores indicative of greater medication adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Harding Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill K, Mann L, Laws KR, Stephenson CM, Nimmo-Smith I, McKenna PJ. Hypofrontality in schizophrenia: a meta-analysis of functional imaging studies. Acta Psychiatr Scand. 2004 Oct;110(4):243-56. doi: 10.1111/j.1600-0447.2004.00376.x. PMID 15352925
- [Background] Karry R, Klein E, Ben Shachar D. Mitochondrial complex I subunits expression is altered in schizophrenia: a postmortem study. Biol Psychiatry. 2004 Apr 1;55(7):676-84. doi: 10.1016/j.biopsych.2003.12.012. PMID 15038995
- [Background] Kann O, Kovacs R. Mitochondria and neuronal activity. Am J Physiol Cell Physiol. 2007 Feb;292(2):C641-57. doi: 10.1152/ajpcell.00222.2006. Epub 2006 Nov 8. PMID 17092996
- [Background] Bloch Y, Applebaum J, Osher Y, Amar S, Azab AN, Agam G, Belmaker RH, Bersudsky Y. Normobaric hyperoxia treatment of schizophrenia. J Clin Psychopharmacol. 2012 Aug;32(4):525-30. doi: 10.1097/JCP.0b013e31825d70b8. PMID 22722511
- [Background] First, M.B., et al., Structured Clinical Interview for DSM-5-Research Version2015, Arlington, VA: American Psychiatric Association.
- [Background] Perkins DO, Leserman J, Jarskog LF, Graham K, Kazmer J, Lieberman JA. Characterizing and dating the onset of symptoms in psychotic illness: the Symptom Onset in Schizophrenia (SOS) inventory. Schizophr Res. 2000 Jul 7;44(1):1-10. doi: 10.1016/s0920-9964(99)00161-9. PMID 10867307
- [Background] Wilkinson, G.S. and G.J. Robertson, Wide Range Achievement Test (WRAT4)2006, Lutz, FL: PAR, Inc.
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] AARC. AARC clinical practice guideline. Oxygen therapy in the home or alternate site health care facility--2007 revision & update. Respir Care. 2007 Aug;52(8):1063-8. No abstract available. PMID 17715561
- [Background] Schizophrenia Spectrum and Other Psychotic Disorders, in DSM-5® Clinical Cases.
- [Background] Auther, A., C. Smith, and B. Cornblatt, Global Functioning: Social Scale (GF: Social). Glen Oaks, NY: Zucker-Hillside Hospital, 2006.
- [Background] Niendam, T., et al., Global Functioning: Role Scale (GF: Role). Los Angeles, CA: University of California, Los Angeles, 2006.
- [Background] Rosenheck RA, Leslie DL, Sindelar J, Miller EA, Lin H, Stroup TS, McEvoy J, Davis SM, Keefe RS, Swartz M, Perkins DO, Hsiao JK, Lieberman J; CATIE Study Investigators. Cost-effectiveness of second-generation antipsychotics and perphenazine in a randomized trial of treatment for chronic schizophrenia. Am J Psychiatry. 2006 Dec;163(12):2080-9. doi: 10.1176/ajp.2006.163.12.2080. PMID 17151158
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Thompson K, Kulkarni J, Sergejew AA. Reliability and validity of a new Medication Adherence Rating Scale (MARS) for the psychoses. Schizophr Res. 2000 May 5;42(3):241-7. doi: 10.1016/s0920-9964(99)00130-9. PMID 10785582
- [Background] Hays, R.D., S. Prince-Embury, and H.Y. Chen, RAND-36 Health Status Inventory1998, San Antonio, TX: The Psychological Corporation.
- [Background] Levine J, Schooler NR. SAFTEE: a technique for the systematic assessment of side effects in clinical trials. Psychopharmacol Bull. 1986;22(2):343-81. No abstract available. PMID 3774930
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Palmer BA, Pankratz VS, Bostwick JM. The lifetime risk of suicide in schizophrenia: a reexamination. Arch Gen Psychiatry. 2005 Mar;62(3):247-53. doi: 10.1001/archpsyc.62.3.247. PMID 15753237